CLINICAL TRIAL: NCT04052893
Title: Postoperative Disease-free Survival and Quality of Life After Modified Radical Mastectomy Versus Expanded Mckissock Surgery for Extensive Intraductal Carcinoma of the Breast: a Prospective Cohort Study Protocol
Brief Title: DFS and QOL After Modified Radical Mastectomy vs. Expanded Mckissock Surgery for EIC of the Breast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Jianyi Li, Principal Investigator, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shengjing-LJY02
Record Dates: First submitted 2019-08-06; First posted 2019-08-12 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms
Keywords: Surgery; Plastic
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Modified Radical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): 100 patients will be assigned into a study group.
  Interventions: Procedure: Expanded Mckissock surgery
- Control group (Active Comparator): 100 patients will be assigned into a control group.
  Interventions: Procedure: Modified radical mastectomy

INTERVENTIONS:
Procedure: Expanded Mckissock surgery — Expanded Mckissock surgery: (1) According to patient's preoperative imaging results and subjective expectations of their own breast morphology, the incision design and breast surface marking will be performed under the standing position. (2) After general anesthesia, the upper limbs will be abducted, and the upper body will be tilted by 15°-20° to dermatize the labeled skin around and below the areola. (3) The medial and lateral flaps will be dissociated to remove the total gland with nipple and areola preserved. (4) The cutting-edge of nipple-areola complex will be sent for cancer screening. The axillary lymph node biopsy or cleaning will be performed along the outer edge of the pectoralis major muscle. (5) The vertical subcutaneous pedicle flaps will be W-folded, and the flaps on both sides will be pulled to the vertical pedicle to reshape the breast. During this process, the breast and armpit drainage tubes will be indwelled.
  Arms: Study group
Procedure: Modified radical mastectomy — The patients will be placed in the supine position. After intravenous anesthesia, the tumor boundary will be marked and the breast will be removed. The vertical subcutaneous pedicle flaps will be W-folded, and the flaps on both sides will be pulled to the vertical pedicle to reshape the breast. During this process, the breast and armpit drainage tubes will be indwelled.
  Arms: Control group

SUMMARY:
Extensive intraductal carcinoma of the breast refers to a type of breast cancer in which ≥ 25% of ductal carcinoma in situ is present in invasive tumors and there is a scattered distribution of ductal carcinoma in situ (DCIS) in or around the invasive carcinoma. Compared with DCIS negative for extensive intraductal component, DCIS positive for extensive intraductal component is not sensitive to radiotherapy. Mckissock surgery was applied in breast-conserving surgery for breast cancer in 2016. Jianyi Li and the team members (Shengjing Hospital of China Medical University, Shenyang, China) applied this technique in breast-conserving surgery with preservation of the nipple-areola complex. This surgical technique is suitable for low-grade malignant tumors and has better prognosis than radical mastectomy. The purpose of this study is to investigate postoperative disease-free survival and quality of life after modified radical mastectomy versus expanded Mckissock surgery for extensive intraductal carcinoma of the breast. Results from this study will indicate the efficacy of expanded Mckissock surgery in the treatment of extensive intraducatal carcinoma of the breast.

DETAILED DESCRIPTION:
Extensive intraductal carcinoma of the breast refers to a type of breast cancer in which ≥ 25% of ductal carcinoma in situ is present in invasive tumors and there is a scattered distribution of ductal carcinoma in situ (DCIS) in or around the invasive carcinoma. Studies have shown that patients with DCIS positive for extensive intraductal component have more residual tumors than patients with DCIS negative for extensive intraductal component. There are still many subclinical tumors in the residual mammary gland after removal of the main invasive tumor foci. This provides the condition for tumor recurrence after breast-conserving surgery, and the risk of tumor recurrence in DCIS positive for extensive intraductal component is 2.52 times that in DCIS negative for extensive intraductal component. Compared with DCIS negative for extensive intraductal component, DCIS positive for extensive intraductal component is not sensitive to radiotherapy.

Mckissock surgery is originated from a breast reduction surgery developed by American doctors in 1970, which can remove glands to the maximum extent. This technique was applied to breast-conserving surgery in 2016, which initiated the application of this operation in malignant tumors. Jianyi Li and the team members (Shengjing Hospital of China Medical University, Shenyang, China) first applied expanded Mckissock surgery in breast-conserving surgery with the nipple-areola complex preserved. This surgical technique is suitable for low-grade malignant tumors. This surgical technique has been performed in 30 patients and results showed that the expanded Mckissock surgery has better prognosis than radical mastectomy. Therefore, this prospective cohort study will compare the postoperative disease-free survival and quality of life between modified radical mastectomy and expanded Mckissock surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with extensive intraductal carcinoma confirmed by hollow needle biopsy;
* the lesion not involving the nipple as confirmed by enhanced MR imaging of the breast;
* Bra cup size: B or higher;
* postmenopausal patients;
* provision of written informed consent.

Exclusion Criteria:

* The cutting edge of nipple-areola complex tested positive for extensive intraductal carcinoma twice;
* preoperative nipple hemorrhage;
* bilateral breast cancer;
* inflammatory breast cancer;
* distant metastasis;
* other cancers or those who receive chest radiotherapy.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival. | 5 years
  Disease-free survival refers to the time from surgical resection of breast cancer to clinically confirmed local recurrence, distant metastasis, second primary tumor diagnosis, or patient death.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer (EORTC) Breast Cancer-Specific Quality of Life Questionnaire (QLQ-BR23) scale | 5 years
  The QLQ-BR23 scale will evaluate the quality of life. The QLQ-BR23 scale consists of 23 items with a full score of 92. Higher score indicates poor quality of life.
Breast symmetry | 5 years
  The symmetry of reconstructed breast will be evaluated using Harris score. The Harris score was described by Harris et al. (Int J Radiat Oncol Biol Phys 1979; 5: 257- 261.) It will be divided into four levels: excellent, good, fair, and poor.
Medical cost | During hospitalization, an average of 2 weeks
  Including medical insurance and commercial insurance reimbursement.

CONTACTS AND LOCATIONS:
Overall Officials: Jianyi Li, Principal Investigator — Shengjing Hospital
Locations (3):
- China (3):
  - General Hospital of Benxi Iron & Steel Industry Group of Liaoning Health Industry Group, Benxi, Liaoning
  - Cancer Hospital of China Medical University, Liaoning Cancer Hospital and Institute, Shengyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning